CLINICAL TRIAL: NCT04880642
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase 3, Multicenter Trial Investigating the Efficacy and Safety of C21 as add-on to Standard of Care in Adult Subjects With COVID-19
Brief Title: A Trial to Investigate Recovery From COVID-19 With C21 in Adult Subjects
Acronym: ATTRACT-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-C21-008; 2021-000264-29 (EudraCT Number)
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — compound 21

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- C21 (Experimental): 50 mg capsules, oral administration twice daily,for 14 days
  Interventions: Drug: C21
- Placebo (Placebo Comparator): placebo capsules, oral administration twice daily,for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C21 — C21
  Arms: C21
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This trial is a randomized, double-blind, placebo-controlled, parallel-group, 2-arm, multicenter trial to evaluate the efficacy and safety of C21 versus placebo as add-on to standard of care (SoC) in adult subjects with COVID-19.

The trial planned to enroll a total of maximum 300 randomized subjects, 150 per arm (oral C21 100 mg twice a day (BID) or placebo for 14 days) according to the 1:1 randomization.

DETAILED DESCRIPTION:
The trial consists of 3 consecutive periods: a screening period of up to 48 hours, a 2-week investigational medicinal product (IMP) treatment period and a follow-up period of up to 7 weeks after last IMP intake.

All subjects went through a series of efficacy, safety, and laboratory assessments. Safety laboratory tests and samples for future exploratory analysis were obtained at the screening visit.

The trial duration for an individual subject was not exceeded 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years or the legal age of consent in the jurisdiction in which the trial was taking place at the time of signing the informed consent (Specific for India; Age ≥18 to ≤65 years at the time of signing the informed consent)
2. Hospitalized due to SARS-CoV-2 infection confirmed by a hospital-approved polymerase chain reaction (PCR) test, documented by either of the following:

   1. PCR positive in sample collected <72 hours prior to randomization (Visit 2); OR
   2. PCR positive in sample collected ≥72 hours and ≤7 days prior to randomization, documented inability to obtain a repeat sample AND progressive disease suggestive of ongoing SARS-CoV-2 infection
3. A score of 5 or 6 on the 8-point ordinal scale:

   1. Score 5: Hospitalized, requiring supplemental oxygen
   2. Score 6: Hospitalized, on non-invasive ventilation or high-flow oxygen device
4. Contraceptive use by men and women of childbearing potential consistent with local regulations regarding the methods of contraception for those participating in clinical studies and according to Appendix 3 in the Protocol (see Section 10.3)
5. Written informed consent, consistent with International Council for Harmonization Good Clinical Practice Revision 2 and local laws, obtained before the initiation of any trial-related procedure
6. Capable of giving signed informed consent as described in Appendix 1 in the Protocol (see Section 10.1.3) which includes compliance with the requirements and restrictions listed in the informed consent form and in this Protocol

   Country specific:
7. Specific for India: For subjects with an ordinal scale score of 5, moderate to severe COVID-19 disease confirmed by at an SpO2≤93 % or a respiratory rate≥24/min on room air. Note: If a subject was on supplemental oxygen with SpO2>93% and respiratory rate<24/min, but desaturation to ≤93 % or increase of respiratory rate to ≥24/min on lower supplemental oxygen or room air is documented during screening, the inclusion criterion was considered to be met.

Exclusion Criteria:

1. Concurrent serious medical condition which in the opinion of the investigator constituted a risk or a contraindication for the participation in the trial or that could interfere with the trial objectives, conduct or evaluation
2. Known, active tuberculosis, active hepatitis B, C, or human immunodeficiency virus (HIV) infection (i.e., HIV with a CD4 count<500 cells/mm³).
3. Moderate or severe impairment of hepatic function (e.g., Child-Pugh class B or C where alterations in the score components were not due to another underlying disease (see Section 8.4.5 in the Protocol)).
4. Severe renal impairment (i.e., estimated glomerular filtration rate (eGFR)≤30 ml/min/1.73m2)
5. COVID-19 symptom onset >21 days prior to screening (Visit 1).
6. Hospitalized due to COVID-19 for >72 hours at screening (Visit 1).
7. Invasive mechanical ventilation or ECMO within 72 hours of screening (Visit 1).
8. Expected need for invasive mechanical ventilation or ECMO in <48 hours in the opinion of the investigator
9. Moderate to severe ARDS (e.g., same-day PaO2/FiO2 ≤200 mmHg; or SpO2/FiO2 ≤232 if arterial blood gas test is not available), if on non-invasive mechanical ventilation or high-flow oxygen.
10. Pregnant or breast-feeding female subjects
11. Any previous and concurrent experimental treatment for COVID-19 that was not considered local SoC.
12. Treatment with the medications listed below within 1 week prior to screening (Visit 1) or anticipated need for such medication during the participation in this trial:

    1. Strong Cytochrome P450 (CYP) 3A4 inducers.
    2. P-glycoprotein (P-gp) substrates with narrow therapeutic index.
    3. High dose Breast Cancer Resistance Protein (BCRP) sensitive substrates.
    4. Warfarin.
    5. Sulphasalazine or rosuvastatin.
13. Current or previous participation in any other clinical trial where the subject had received a dose of IMP within 1 month or 5 half-lives of the IMP, whichever was longest, prior to screening (Visit 1).
14. Positive pregnancy test (see Section 8.4.6 in the Protocol).
15. Abnormal laboratory value at screening (Visit 1) indicating a potential risk for the subject if enrolled in the trial as evaluated by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Horton, MD, Principal Investigator — Johns Hopkins University School of Medicine, Baltimore, USA
Locations (60):
- United States (6):
  - University of California Irvine Medical Center, Orange, California
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Parkview Physicians Group - Infectious Diseases, Fort Wayne, Indiana
  - Trinity Health, Minot, North Dakota
  - Lehigh Valley Hospital - 17th Street, Allentown, Pennsylvania
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
- Argentina (4):
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Hospital Italiano Rosario - Centro, Rosario, Santa Fe Province
  - Hospital Italiano Rosario, Rosario, Santa Fe Province
  - Nuevo Hospital San Roque, Córdoba
- Brazil (7):
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu
  - Hospital Brasília, Brasília
  - Fundação Universidade de Caxias do Sul, Caxias do Sul
  - Centro de Pesquisas Clínicas de Natal, Natal
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital Alemão Oswaldo Cruz - Paulista, São Paulo
- Colombia (3):
  - Clinica Somer, Rionegro, Antioquia
  - Fundación Santa Fe de Bogotá, Bogotá, Cundinamarca
  - Hospital Universitario San Ignacio, Bogotá, Cundinamarca
- Czechia (4):
  - Fakultní Nemocnice u sv. Anny v Brně II. Interní Klinika kardiologická JIP,, Brno, South Moravian
  - Fakultní Nemocnice u sv. Anny v Brne Number 1, Brno
  - Nemocnice Slaný, Slaný
  - Masarykova nemocnice v Ústí nad Labem, Ústí nad Labem
- India (13):
  - Chettinad Hospital and Research Institute, Mahabalipuram, Chennai
  - Civil Hospital and B J Medical College, Ahmedabad, Gujarat
  - Smt. Kashibai Navale Medical College and General Hospital, Pune, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Malabar Medical College Hospital and Research Centre, Kozhikode, Kerala
  - Elite Mission Hospital, Thrissur, Kerala
  - Chirayu Medical College and Hospital, Bhopal, Madhya Pradesh
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - Meditrina Institute of Medical Sciences, Nagpur, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Rajiv Gandhi Medical College, Thane, Maharashtra
  - Jawaharlal Nehru Institute of Medical Sciences, Imphal, Manipur
- Philippines (7):
  - The Medical City, Iloilo City, Iloilo
  - St. Luke's Medical Center - Global City, City of Taguig
  - Southern Philippines Medical Center, Davao City
  - West Visayas State University Medical Center, Iloilo City
  - Makati Medical Center, Makati
  - Lung Center of the Philippines, Quezon City
  - Quirino Memorial Medical Center, Quezon City
- Russia (5):
  - Clinical Infectious Disease Hospital 1 of the Moscow Department of Health, Moscow
  - Alexandrovskaya State Hospital, Saint Petersburg
  - Nikolaevskaya State Hospital, Saint Petersburg
  - Pokrovskaya City Hospital, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution City Hospital Number 40 of the Kurortny District, Saint Petersburg
- South Africa (3):
  - Mediclinic Southern Africa, Tongaat, KwaZulu-Natal
  - TASK Eden, George, Western Cape
  - Tygerberg Hospital, Tygerberg Hills, Western Cape
- Ukraine (8):
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhia, Zaporizhzhia Oblast
  - City Clinical Hospital №6 of the Dnipro City Council, Dnipro
  - City Clinical Hospital №13" Of Kharkiv City Council, Kharkiv
  - Regional Clinical Hospital of Infectious Diseases, Kharkiv
  - Kyiv city clinical hospital number 12, Kiev
  - Oleksandrivska Kyiv City Clinical Hospital, Kyiv
  - Vinnytsia City Clinical Hospital №1, Vinnytsia
  - Hospital №1 of Zhytomyr City Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 316 subjects were screened. Of those, 44 subjects were screening failures, 39 for failure to meet eligibility criteria, 3 due to withdrawal by the subject, and 2 for other reasons. The remaining 272 subjects were randomized. 5 of the randomized subjects did not receive treatment.
  The screening period was from signing of ICF until randomization.
Groups:
- C21 Treatment: Oral C21 treatment 100 mg twice daily for 14 days.
- Placebo Treatment: Oral placebo treatment twice daily for 14 days.
Period: Randomization
Arm/Group | C21 Treatment | Placebo Treatment
Started | 136 | 136
Completed | 134 | 133
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3
Period: Treatment Period
Arm/Group | C21 Treatment | Placebo Treatment
Started | 134 | 133
Completed | 122 | 121
Not Completed | 12 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Death | 6 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Discontinuation criteria of eGFR | 0 | 1
Period: Follow-up
Arm/Group | C21 Treatment | Placebo Treatment
Started (A total of 8 subjects (5 subjects in the C21 group and 3 subjects in the placebo group) discontinued treatment but continued to participate in the trial.) | 122 | 121
Completed | 117 | 118
Not Completed | 5 | 3
Not completed — Death | 4 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C21 Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [18 to 79] | 56.5 [21 to 91] | 55.0 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 120
  Male | 79 | 73 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 127 | 127 | 254
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 43 | 45 | 88
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 90 | 87 | 177
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Colombia | 2 | 0 | 2
  United States | 4 | 4 | 8
  Czechia | 20 | 19 | 39
  Philippines | 3 | 5 | 8
  Ukraine | 54 | 55 | 109
  Brazil | 4 | 5 | 9
  South Africa | 2 | 3 | 5
  India | 38 | 38 | 76
  Russia | 9 | 7 | 16
Height [Mean (Full Range); unit: Cm] | 168.8 [145 to 195] | 167.6 [149 to 187] | 168.2 [145 to 195]
Weight [Mean (Full Range); unit: Kg] | 81.89 [50.0 to 200.0] | 79.26 [43.0 to 159.0] | 80.58 [43.0 to 200.0]
Body mass index [Mean (Full Range); unit: Kg/m^2] | 28.71 [19.0 to 69.2] | 28.14 [13.3 to 57.0] | 28.42 [13.3 to 69.2]

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality up to Day 60
Description: Proportion of subjects in the mITT (all randomised, including 5 subjects not treated) with death up to Day 60 follow-up
Time Frame: Day 1 to Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 136 | 136
Participants
  Death | 10 | 10
  Censored | 126 | 126
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Superiority — The null hypothesis was that the there was no difference in survival up to Day 60 between the two groups and was to be rejected in favour of the alternative hypothesis i.e. a difference in survival up to Day 60 between the two groups excisted. The overall 2-sided significance level of 5% was applied to the primary endpoint; p = 0.949, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.40 to 2.36]

2. Secondary Outcome: Time to Sustained Hospital Discharge up to Day 60
Description: Time to sustained hospital discharge from Day 1 to Day 60: Time to sustained hospital discharge was defined as the time to the date of discharge from the initial hospitalization or re-hospitalization due to COVID-19 after which the subject was not re-hospitalized for COVID-19 related reasons.
Time Frame: Day 1 to Day 60
Population: ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 136 | 136
Days | 9.0 [7.0 to 11.0] | 9.0 [8.0 to 11.0]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Superiority; p = 0.301, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.91 to 1.52]

3. Secondary Outcome: Supplemental Oxygen-free Days up to Day 29
Description: Supplemental oxygen-free days from Day 1 up to Day 29, observed range 0 to 28 days. Subjects with deaths imputed as -1 day according to SAP and FDA guidance. Outcome was identical in both groups for both median and range
Time Frame: Day 1 to Day 29, maximum 28 Days
Population: ITT
Measure: Median (Full Range); unit: Days
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 136 | 136
Days | 23.0 [-1 to 28] | 23.0 [-1 to 28]
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Superiority; p = 0.425, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-1 to 1]

4. Secondary Outcome: Proportion of Subjects Free of Respiratory Failure, Defined as an 8-point Ordinal Scale Score ≤5, at Day 15
Description: Proportion of subjects free of respiratory failure, defined as an 8-point ordinal scale score ≤5, at Day 15. Missing data imputed by MI, proportion given are average over the imputations.
Time Frame: Day 15
Population: ITT
Measure: Number; unit: proportion of responders
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 136 | 136
proportion of responders | 0.884 | 0.901
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Superiority; p = 0.671, Regression, Logistic; Risk Difference (RD) = -1.7, 95% CI 2-sided [-9.3 to 6.0], Standard Error of Mean 3.91

5. Secondary Outcome: Proportion of Subjects Discharged From Hospital and Free of Supplemental Oxygen at Day 15
Description: Proportion of subjects discharged from hospital and free of supplemental oxygen at Day 15. Missing data imputed by MI, proportion given are average over the imputations.
Time Frame: Day 15
Population: ITT
Measure: Number; unit: proportion of responders
Arm/Group | C21 Treatment | Placebo Treatment
Number analyzed (Participants) | 136 | 136
proportion of responders | 0.676 | 0.679
Statistical Analysis 1: Comparison: C21 Treatment vs Placebo Treatment; Test type: Superiority; p = 0.948, Regression, Logistic; Risk Difference (RD) = -0.4, 95% CI 2-sided [-11.4 to 10.6], Standard Error of Mean 5.62

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing of informed consent until day 29 (visit 31 in the follow-up period). Serious adverse events were collected from signing of informed consent until day 60 (visit 32 in the follow-up period). Adverse events occurring after the first Investigational Medical Product (IMP) intake were considered treatment-emergent adverse events (TEAEs) in the statistical analysis.
Description: All-Cause Mortality was monitored in all randomized subjects (n=272) whereas Serious and Other Adverse Events were assessed in the safety population including treated subjects only (n=267). 5 randomized subjects, but not treated, were not included in the evaluation of adverse events. None of these 5 subjects had any reported adverse events and thereby no deaths.
Arm/Group | C21 Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 10/136 | 10/136
Serious Adverse Events (participants affected / at risk) | 15/134 | 13/133
Other Adverse Events (participants affected / at risk) | 22/134 | 24/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 Treatment (N=134) | Placebo Treatment (N=133)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Frederick's syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 Treatment (N=134) | Placebo Treatment (N=133)
Alanine aminotransferase increased (Investigations) | 7 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (7)
Pyrexia (General disorders) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 4 (4) | 5 (6)
Asthenia (General disorders) | 4 (4) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT04880642/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT04880642/SAP_001.pdf